CLINICAL TRIAL: NCT07313631
Title: Women's Insurance for State Health - An Impact Evaluation of Health Insurance Provided Under the Basic Health Care Provision Fund in Taraba State, Nigeria
Brief Title: Impact Evaluation of Access to Free Low-Cost Health Insurance in Nigeria's Taraba State
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NFWP_Taraba_HealthInsurance
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Health Behavior; Economic Problems; Health Status; Healthcare Utilization
Keywords: Health insurance; Care-seeking behavior; Healthcare utilization; Nigeria
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial at the Women Affinity Group (WAG) level; 1,000 WAGs randomly assigned (stratified by ward and age strata) into treatment or control (500 each), with four women sampled per group (4,000 total participants).
Who Masked: Outcomes Assessor
Masking Description: The survey enumerators will not blinded to the treatment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Health insurance offer) (Experimental): Randomly-selected members of selected Women Affinity Groups (WAGs) randomized to the treatment arm receive an offer for a free, 12-month health insurance policy under the Taraba State Health Insurance Agency's Basic Minimum Package of Health Services (BMPHS), covering essential primary and secondary care (including consultations, preventive services, maternal and child health, emergency care, mental health, and laboratory services).
  Interventions: Other: No-Cost Health Insurance
- Control (No insurance offer) (No Intervention): Members of WAGs randomized to the control arm do not receive the insurance coverage offer during the study period and continued with usual access to care without project-provided coverage.

INTERVENTIONS:
Other: No-Cost Health Insurance — Provision of a free, 12-month insurance policy from the Taraba State Health Insurance Agency that covers the Basic Minimum Package of Health Services (BMPHS), including outpatient and inpatient consultations, preventive and reproductive health services, maternal and child health care, mental health care, emergency services, and laboratory testing.
  Arms: Treatment (Health insurance offer)

SUMMARY:
The objective of this study is to examine the impact of a free health insurance offer on healthcare use, spending, self-reported health, and economic participation of women in Taraba state of Nigeria.

DETAILED DESCRIPTION:
This study aims to evaluate a health-insurance intervention implemented under the World Bank-funded Nigeria for Women Project (NFWP) in Taraba State. Women in Women Affinity Groups (WAGs) received an offer for a free, 12-month policy under the Taraba State Health Insurance Agency's Basic Minimum Package of Health Services (BMPHS), which covers essential primary and secondary care, including consultations, preventive services, maternal and child health, mental health, emergency care, and laboratory services, normally priced at ₦12,000 annually. We are using a randomized controlled trial design in Bali Local Government Area (LGA). Using administrative data on WAG enrollment, we randomly assigned 1,000 WAGs (stratified by ward and mean participant age) to either treatment (n=500) or control (n=500). Within each WAG, four women were randomly selected to enroll in the study, yielding 4,000 participants (2,000 insured; 2,000 controls). The study focuses on outcomes related to healthcare utilization, health status, out-of-pocket expenditures, and women's economic participation. The findings are expected to inform policy on expanding health insurance coverage as a strategy to improve women's health and promote their economic empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Members of one of 1,000 randomly selected women's groups operating in Bali local government area in Taraba State, Nigeria.

Exclusion Criteria:

* At least 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Respondent has health insurance | 6 months, 9 months, 11 months post treatment.
  Zero if not no health insurance, 1 if has health insurance.
Has health insurance card | 6 months, 9 months, 11 months post treatment
  Zero if respondent has no health insurance card, 1 if they have a health insurance card.
Respondent has successfully used health insurance for consultations, diagnoses, medications, or tests. | 6 months, 9 months, 11 months.
  Zero if respondent has not successfully used health insurance for consultations, diagnoses, medications, or tests. 1 if the respondent has successfully used health insurance for consultations, diagnoses, medications, or tests.
Sought treatment for most recent illness | 6 months, 9 months, 11 months.
  Zero if respondent did not seek care for most recent illness. 1 if respondent did seek care for most recent illness
Number of health facility visits in last 3 months. | 6 months, 9 months, 11 months.
  Reported number of health facility visits outside the home in the last 3 months.
Most recent health facility visit was to a public sector facility | 6 months, 9 months, 11 months.
  Zero if last care event was in a private facility, 1 if last care seeking event was in a public facility
Money for health care is a key barrier | 6 months, 9 months, 11 months.
  Zero if "getting money needed for advice or treatment" is not listed as a barrier. 1 if "getting money needed for advice or treatment" listed as a barrier.
Most recent birth was in a health facility | 6 months, 9 months, 11 months.
  Zero if most recent birth was not in a government or private health facility. 1if most recent birth was in a government or private health facility. Limited to births in last 3 months.
Child has received any vaccinations | 6 months, 9 months, 11 months.
  Zero if children aged under 12 months has not received any vaccinations. 1 if child has received at least one vaccination.
Total cost of most recent healthcare | 6 months, 9 months, 11 months.
  Total cost of most recent healthcare visit, winsorized at the 1% and 99% levels.
Most recent care episode reflects catastrophic health expenditure | 6 months, 9 months, 11 months.
  1 if most recent healthcare visit expenditure represents represents greater than 10% of household consumption
Total indebtedness from healthcare or illness-related expenses | 6 months, 9 months, 11 months.
  Total amount of money owed for medical expenses, winsorized at the 1% and 99% levels.
Respondent is depressed | 6 month, 9 month, 11 month.
  Score equal to or greater than 10 on Center for Epidemiologic Studies Depression Scale.
Perceived health status | 6 months, 9 months, 11 months.
  Response to the following question: Think about your health over the last 3 months, including any long-term illnesses, hospital or clinic visits, or other ailments, how would you rate your health on a scale of 1-10 where 1 is very low health and 10 is very healthy with no ailments?
Number of productive days lost to severe illness in the past 3 months | 6 months, 9 months, 11 months
  Reported number of productive days lost to severe illness in the past 3 months

SECONDARY OUTCOMES:
Has ever tried to use health insurance | 6 months, 9 months, 11 months post treatment
  Zero if respondent has never tried to use health insurance, 1 if respondent has tried to use health insurance
Number of antenatal care visits | 6 months, 9 months, 11 months.
  Number of antenatal care visits for any births in last 3 months
Most recent health facility care event visit was to a secondary/tertiary care facility (hospital) | 6 months, 9 months, 11 months.
  1 if most recent health facility care event visit was to a secondary/tertiary care facility (hospital). 0 if visit was to a primary care facility or informal care facility.
Received lab test as part of antenatal care in most recent pregnancy | 6 months, 9 months, 11 months.
  1 if received any lab tests as part of antenatal care in most recent pregnancy from births in last year. 0 otherwise.
Child has received OPV | 6 months, 9 months, 11 months.
  1 if child born in last 12 months and age-eligible for OPV vaccine has received it. 0 if child born in last 12 months and age-eligible for OPV vaccine but has not received it.
Child has received BCG vaccine | 6 months, 9 months, 11 months.
  1 if child born in last 12 months and age-eligible for BCG vaccine has received it. 0 if child born in last 12 months and age-eligible for BCG vaccine but has not received it.
Child has received measles vaccine | 6 months, 9 months, 11 months.
  1 if child born in last 12 months and age-eligible for measles vaccine has received it. 0 if child born in last 12 months and age-eligible for measles vaccine but has not received it.
Economically active in the last 7 days | 6 months, 9 months, 11 months.
  1 if respondent reports working, either paid or unpaid, in the last 7 days. This includes: work as an employee for a wage, salary, commission or any payment in kind; running a non-farm business; help in any kind of nonfarm business; work on your own farm or household agricultural activities; and unpaid apprentice work.
  0 if no work in the last 7 days.
Hours engaged in economic activities in the last 30 days | 6 months, 9 months, 11 months.
  Total number of hours reported towards economic activities in the last 30 days. Calculated as days worked in a given activity times hours spent in a given activity, summed over activities.
Total income over past 30 days. | 6 months, 9 months, 11 months.
  Reported income from all economic activities over the last 30 days, winsorized at the 1% and 99% levels.
Total value of current savings | 6 months, 9 months, and 11 months post treatment.
  Total value of current savings, winsorized at the 1% and 99% levels.
Total value of current borrowing | 6 months, 9 months, and 11 months post treatment.
  Value of all outstanding borrowing owed for food, medical expenses, loans, social occasions, school fees, businesses, and other. Winsorized at the 1% and 99% levels.
Household decision making | 6 months, 9 months, and 11 months post treatment.
  1 if the respondent feels she has input into most or all household decisions, 0 if she has input into none, few, or some decisions.
Respondent makes decisions about savings | 6 months, 9 months, 11 months post treatment.
  1 if respondent can make their own personal decisions regarding savings (at least to a small extent). 0 if respondent can not make their own personal decisions regarding savings
Health insurance knowledge | 6 months, 9 months, 11 months.
  Number of questions correct about what health insurance does/does not cover:
  Health insurance covers the registration fee at a health facility. Health insurance covers the consultation fee you pay to see a doctor or nurse. Health insurance covers the cost of laboratory tests. Health insurance covers the cost of medicines or drugs. Health insurance covers the cost of treatment.
Trust in state government | 6 months, 9 months, 11 months post treatment
  1 if respondent has trusts state government (a great deal of trust or trust somewhat), 0 if no trust at all or trust just a little.
Trust in local government authority | 6 months, 9 months, and 11 months post treatment.
  1 if respondent has trusts local government authority (a great deal of trust or trust somewhat), 0 if no trust at all or trust just a little.

CONTACTS AND LOCATIONS:
Locations (1):
- Bali LGA, Beli, Taraba State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified dataset with all collected IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We will release data two years after each data collection:
  Round 1: November 2027 Round 2: February 2028 Round 3: April 2028
Access Criteria: The data will be publicly available on the World Bank's microdata website. Use of the dataset must be acknowledged using a citation which would include:
  1. the identification of the Principal Investigators,
  2. the title of the survey (including country, acronym and year of implementation)
  3. the survey reference number
  4. the source and date of download